CLINICAL TRIAL: NCT02308800
Title: Negative Pressure Wound Therapy as a Drug Delivery System
Brief Title: Negative Pressure Wound Therapy as a Drug Delivery System (ADANPWT)
Acronym: ADA NPWT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 092014-016
Record Dates: First submitted 2014-11-07; First posted 2014-12-04 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Foot Ulcer, Diabetic
Keywords: diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quantum™ Therapy/NPWT with Prontosan (Active Comparator): Quantum™ Negative Pressure Wound Therapy with Prontosan irrigant.
  Interventions: Device: Quantum™ Therapy - NPWT with Prontosan
- Quantum™ Therapy (Active Comparator): Quantum™ Negative Pressure Wound Therapy without irrigant.
  Interventions: Device: Quantum™ Therapy

INTERVENTIONS:
Device: Quantum™ Therapy - NPWT with Prontosan — Negative pressure wound therapy with Prontosan irrigation.
  Arms: Quantum™ Therapy/NPWT with Prontosan
Device: Quantum™ Therapy — Negative pressure wound therapy without irrigation.
  Arms: Quantum™ Therapy

SUMMARY:
The investigators plan a randomized clinical trial of 150 patients with infected diabetes-related lower extremity wounds to compare the clinical and economic effectiveness of negative pressure wound therapy with continuous irrigation and negative pressure wound therapy without irrigation.

The investigators will enroll 150 patients from two centers: The University of Texas Southwestern University Hospital and Parkland Hospital. The investigators will screen and enroll patients with wounds in the inpatient setting. Patients will randomized to receive traditional NPWT or NPWT with continuous irrigation while they are hospitalized. The average hospitalization for patents that receive NPWT is 13.3 days. Patients that do not have their wound surgically closed during hospitalization will be discharged with negative pressure wound therapy without irrigation for up to a total of four weeks of therapy. After discharge from the hospital, subjects will be seen twice weekly by home health, and the investigators will evaluate subjects in clinic every 7 days (±7 days) for a total of 16-week period or until the wound heals.

DETAILED DESCRIPTION:
Screening Procedures

* Review and sign the Informed Consent and HIPAA Authorization
* The study doctor will review the inclusion and exclusion criteria
* Demographics (such as age, gender, race or ethnicity)
* Sitting blood pressure and pulse at admission
* Collection of Height and weight at admission
* Collection of the medical and surgical history
* Collection of the history of the wound
* Wound assessment(s) - wound etiology, wound history, location of study wound and infection assessment
* Hyperspectral imaging within 30 days of screening
* Vascular/Neurological evaluation - we will do various tests and measurements to assess the sensation (feeling) and circulation (blood flow) in the subject's feet and lower legs. To assess the sensation, we will do a monofilament sensory test and a vibration threshold perception test on the study foot. We will calculate the neuropathy disability score of both feet. To assess circulation, we will record Skin Perfusion Pressures in the study foot using a Sensilase System (Vasamed, Eden Prairie, MN) within 30 days of screening. We will calculate the ankle brachial index (ABI) at screening and collect available arterial doppler data from the medical record within 6 months of screening. None of these tests are invasive (using needles), uncomfortable or have risks greater than standard care.
* Results of standard-of-care laboratory tests including a white blood cell count, blood chemistry (tests to see how well organs, such as the liver and kidneys are working), glycated hemoglobin, albumin, prealbumin, erythrocyte sedimentation rate, C-reactive protein and blood glucose. Results of a serum pregnancy test (standard care for women of child-bearing potential as part of pre-op labs) will also be collected. Collection of a list of the subject's current antibiotics
* We will provide the SF-36 Questionnaire and other patient-reported outcomes questionnaires and collect them while subjects are inpatient.

This visit will last about 2 hours.

If you qualify for the study, you will participate in the following procedures:

Group Assignment

If the researchers believe the subject can take part in this study, s/he will be assigned randomly (like a flip of a coin) to receive one of the following therapies:

* Negative Pressure Wound Therapy with Irrigation
* Negative Pressure Wound Therapy without Irrigation

The group is assigned randomly (like flipping a coin). The sponsor or researchers do not know in advance what group assignment each subject will receive. Neither the subject nor the researchers will be allowed to choose which group s/he is assigned to.

Study Intervention

The subject will receive either:

* Quantum™+Simultaneous Irrigation (NPWTi) - Negative Pressure Wound Therapy with Prontosan®, or
* Quantum™(NPWT) -Negative Pressure Wound Therapy (without Prontosan®)

Assigned therapy will continue in the hospital until the physician determines that the wound is ready for closure. If the subject's wound is healing, study therapy will be discontinued and standard dressings will be applied. If surgical closure is needed, the subject will return to the Operating Room for a procedure to close the wound.

If the wound is not ready for closure during the hospital stay, subjects will continue NPWT at home. NPWT at home will be without irrigation.

Procedures and Evaluations during the Research The study therapy will only be given while the subject is in the hospital. If the subject's wound is not ready for closure during the hospital stay, the subject will continue NPWT at home. NPWT at home will be without irrigation. Once the therapy is stopped s/he will continue to be followed by the study doctor. After the subject is released from the hospital s/he will need to see the study doctor during regular post-operative visits. The study doctor will continue to check the wound. If the wound closes, s/he will see the study doctor 30 days later to have the closed wound checked.

Day of First Surgery:

* 3D images after the surgery with eKare Insight device
* Tissue and bone samples - the doctor will take 2 small samples of tissue from the subject's wound before debridement (removal of dead or unhealthy tissue), and after debridement (clean margins) and 1 sample of bone before debridement in case of bone infection, and these tissue samples will be kept and tested for the amount and type of bacteria that are present (qPCR analysis/laboratory analysis).
* Wound measurements after the surgery
* The study doctor will decide if the subject still qualifies to be in the study
* Randomization (like flipping a coin) to either Quantum™ NPWT with Irrigation or Quantum™ NPWT without Irrigation
* Placement of therapy on the wound
* Collection of current antibiotics
* Collection of adverse event information

Daily Treatments (while in the hospital):

* Collection of current antibiotics
* Collection of adverse event information

This will take about 15 minutes.

Additional Surgery (if needed to remove dead tissue or to close the wound):

* Tissue sample - the doctor will take 2 small samples of tissue from the subject's wound after debridement (clean margin), and these tissue samples will be kept and tested for the amount and type of bacteria that are present (qPCR analysis/laboratory analysis)
* 3D images of the wound after the surgery/debridement at bedside with eKare Insight device if the wound is still open
* Wound measurements after the surgery/debridement at bedside
* Wound closure or placement of therapy on the wound
* Collect current antibiotics
* Collect adverse event information

If the subject's wound is not closed upon hospital discharge, NPWT will continue at home without irrigation.

Home Health Visits If the subject continues to receive NPWT after hospital discharge, the subject will be seen twice weekly by a home health nurse for dressing changes. The home health nurse will collect sitting blood pressure and pulse rate. Amount, type and character of drainage will be documented, as well as any adverse events and changes to concomitant medications. Offloading will be reapplied after dressing changes.

Follow-Up Visits per standard of care (after therapy has stopped):

* Dressing change / removal / Offloading
* Wound measurements and infection assessment
* Results of standard-of-care laboratory tests including a white blood cell count, blood chemistry (tests to see how well organs, such as the liver and kidneys are working), glycated hemoglobin, albumin, prealbumin, erythrocyte sedimentation rate, C-reactive protein and blood glucose.
* 3D image of the wound with eKare device (if indicated, if the wound is still open)
* Collection of current antibiotics
* Collection of adverse event information

These visits will take about 30 minutes.

End of Study - Wound Closure Follow-up Visit (30 days +/-7 days after your wound closes, if it closes within 12 weeks from Day of first surgery) or Week 16:

* Closed wound assessment
* For subjects whose wound has not closed:

  3D images of the wound with eKare device Return to standard care
* Collection of current antibiotics
* Collection of adverse event information
* SF-36 Questionnaire and other patient-reported outcomes questionnaires

This visit will take about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Men/women ≥21 years old
* Foot or ankle wounds sized 5 cm2 -100 cm2
* ABI≥0.5 or toe pressures >30 mmHg

Exclusion Criteria:

* Active Charcot arthropathy
* Unable to use NPWT at home
* Untreated bone or soft tissue infection
* Unable to keep research appointments
* Active alcohol or substance abuse (> 14 drinks per week over the last 3 months) or substance abuse (current use of cocaine, heroine or methamphetamine or if drug or alcohol use will interfere with follow up visits in foot clinic in the opinion of the investigator)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Compare clinical outcomes (time to wound healing, number of surgeries) with Negative Pressure Wound Therapy with irrigation and Negative Pressure Wound Therapy without irrigation. | Up to 12 weeks
  The investigators expect that patients treated with NPWT with irrigation will a have higher proportions of wounds that heal, fewer surgeries, and faster wound healing trajectories when compared to patients treated with traditional NPWT without irrigation.

SECONDARY OUTCOMES:
Compare quantitative cultures (bacterial load as measured by qPCR) and number of clinical infections in patients treated with NPWT with irrigation compared to conventional NPWT. | Up to 12 weeks
  The investigators expect that patients treated with NPWT and irrigation will have a significantly lower bacterial load, and fewer and less severe clinical infections.

OTHER OUTCOMES:
Compare responses to the HR-QOL questionnaires of patients treated with NPWT with irrigation compared to conventional NPWT. | Up to 12 weeks
  The investigators expect that patients treated with NPWT and continuous irrigation will have significantly higher indicators of functional health and well-being as compared with standard NPWT

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No